CLINICAL TRIAL: NCT01667991
Title: Evaluation of the American Thoracic Society Criteria for Predicting Multidrug-resistant Bacteria in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Department of Critical Care Medicine, Zhong-Da Hospital, School of Medicine Southeast University, Southeast University, China
Other Study IDs: MDR in China 123
Record Dates: First submitted 2012-08-12; First posted 2012-08-17 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Infection
Keywords: Colonization; infection; multidrug-resistant bacteria; guideline
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Appropriate initial antibiotic treatment based on early diagnosis of etiology will improve the outcome of sepsis. The incidence rates of multidrug-resistant (MDR) bacteria, which are different between countries, will affect the accuracy of etiological diagnoses according to the American Thoracic Society (ATS) guidelines. Therefore the investigators determined the accuracy of the ATS criteria in predicting infection or colonization related to MDR bacteria in China.

DETAILED DESCRIPTION:
All data concerning patient characteristics at ICU admission and during ICU stay were prospectively collected.Screening for MDR bacteria (using nasal swabs, tracheal aspirates from intubated patients and specimens from the infection location) was performed at ICU admission and discharge. Risk factors for infection or colonization with MDR bacteria were recorded, and the accuracy of the ATS criteria in predicting infection or colonization with these bacteria at ICU admission was documented. All of the infected patients were treated by the attending physician, and the choice and adjustment of antibiotic were in accordance with the recommendations of the ATS guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in the ICU were eligible for this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to icu
Sampling Method: Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2010-04; Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Xie, MD, Study Director — Zhongda Hospital

REFERENCES:
- [Derived] Xie J, Ma X, Huang Y, Mo M, Guo F, Yang Y, Qiu H. Value of American Thoracic Society guidelines in predicting infection or colonization with multidrug-resistant organisms in critically ill patients. PLoS One. 2014 Mar 19;9(3):e89687. doi: 10.1371/journal.pone.0089687. eCollection 2014. PMID 24647408